CLINICAL TRIAL: NCT02666872
Title: Evaluation of a New Educational Strategy Promoting Vaccination in Maternity in Quebec Based on Motivational Interviewing Techniques: PROMOVAQ Study
Brief Title: Evaluation of an Intervention PROMOting VAccination in Maternity in Quebec
Acronym: PROMOVAQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: CHU de Quebec-Universite Laval (Other); St. Justine's Hospital (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Arnaud Gagneur, MD, Ph.D, Associate Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-074; 27505 (Other Grant/Funding Number: Fonds de recherche du Québec - Santé (FRQS))
Record Dates: First submitted 2016-01-19; First posted 2016-01-28 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Motivational Interviewing
Keywords: Vaccination; Infant; Parents; Intention
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational interviewing on vaccination (Experimental): An educational strategy based on motivational interviewing of approximately 15 minutes to promote vaccination, in maternity ward.
  Interventions: Behavioral: Motivational interviewing
- Brochure about vaccines for infants (No Intervention): Parents in the control group only received a brochure about vaccines for infants. This brochure is given to all fathers and mothers giving birth to the CHUS, participating or not at our study.

INTERVENTIONS:
Behavioral: Motivational interviewing
  Arms: Motivational interviewing on vaccination

SUMMARY:
Vaccination greatly reduced mortality and morbidity from many preventable diseases. However, to avoid the resurgence of these diseases and the human drama associated, high vaccine coverage should be maintained in the population. Yet in Quebec, vaccine coverage (VC) in young children remains suboptimal, especially caused by a proportion of parents who are ambivalent about the safety and effectiveness of vaccines. In this context, the Provincial Immunization Committee developed in 2010 a Quebec's immunization promotion plan.

Therefore, our research team tested and validated across the Eastern Townships, a vaccination promotion concept by means of an educational intervention within maternities, based on motivational interviewing techniques. This intervention has not only significantly increased the intention of vaccination (+15%) within parents who had received the intervention but also increased their child vaccination coverage (+7.5% at 7 months). This is the purpose of the PROMOVAQ study (PROmotion of VAccination in Quebec) This research project evaluated the impact of an educational strategy based on motivational interviewing techniques within maternity ward on infants' VC. This strategy has been tested through a provincial study (Montreal, Quebec, Sherbrooke) including more than 2500 families.

At term, this research program will offer the Quebec's Health Ministry an optimal strategy for immunization awareness so that Quebec's children may grow healthy and thrive.

ELIGIBILITY:
Inclusion Criteria:

* Parents of all infants born in each participating maternity hospitals
* In Sherbrooke, inclusion limited to parents residing in the region of the Eastern Townships
* In Québec, inclusion limited to parents residing in the National Capital region.

Exclusion Criteria:

* Minor parents
* Parents who do not speak English or French
* Any health condition of the child or the mother needing acute care. That is to say, if the child must be hospitalized in neonatology, or if the mother has an incompatible condition with an interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2719 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Vaccination status of the child at 7 months of age | 10 months
  Data was collected at 10 months of age for all children from regional immunization registries or self-reported by parents over the phone. Vaccination coverage is then defined by the number of infants who received all recommended childhood vaccines at 7 months of age by the total number of children.

SECONDARY OUTCOMES:
Vaccination status of the child at 3 and 5 months of age | 10 months
  Data was collected at 10 months of age for all children from regional immunization registries or self-reported by parents over the phone. Early vaccination coverage is then defined by the number of infants who received all recommended childhood vaccines at 3 and 5 months of age by the total number of children.
Vaccination status of the child at 13, 19 and 24 months of age | 24 months
  Data will be collected at 24 months of age for all children from regional immunization registries or self-reported by parents over the phone. Long-term vaccination coverage is then defined by the number of infants who received all recommended childhood vaccines at 13, 19 and 24 months of age by the total number of children.
Intention's parents to vaccination assessed by a questionnaire based on the Health Belief Model | Within the 20 minutes right before the intervention and within the first 20 minutes right after the intervention
Hesitancy 's parents to vaccination by a questionnaire based on the Opel's tool to measure vaccine hesitancy | Within the 20 minutes right before the intervention and within the first 20 minutes right after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Gagneur, MD, Ph.D, Principal Investigator — Sherbrooke University
Locations (4):
- Canada (4):
  - McGill University Health Centre (Hôpital de Montréal pour enfants), Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
  - CHU de Québec - CHUL, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Derived] Gagneur A, Quach C, Boucher FD, Tapiero B, De Wals P, Farrands A, Lemaitre T, Boulianne N, Sauvageau C, Ouakki M, Gosselin V, Gagnon D, Petit G, Jacques MC, Dube E. Promoting vaccination in the province of Quebec: the PromoVaQ randomized controlled trial protocol. BMC Public Health. 2019 Feb 6;19(1):160. doi: 10.1186/s12889-019-6468-z. PMID 30727991
- See also: Results from PROMOVAC study in Eastern Townships (pilot study before PROMOVAQ) — http://www.santecom.qc.ca/Bibliothequevirtuelle/Estrie/9782981383013.pdf